CLINICAL TRIAL: NCT06497140
Title: A Randomized Sham-controlled, Multicenter Trial on the Effect of Genicular Arteries Embolization in Symptomatic Knee Osteoarthritis
Brief Title: Effect of Genicular Arteries Embolization in Symptomatic Knee Osteoarthritis LipioJoint-2
Acronym: LIPIOJOINT-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP230828; PHRC-22-0033 (Other Grant/Funding Number: French Ministry of Health); 2023-508844-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: Embolization; Pain; Randomized sham-controlled trial
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, multicenter trial comparing GAE using an ethiodized oil-based emulsion with a sham procedure in patients with symptomatic knee osteoarthritis.
  Randomization in a 2:1 ratio of GAE using an ethiodized oil-based emulsion to the sham procedure will be performed with stratification on Kellgren and Lawrence score (2-3 versus 4).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the personal of the Interventional Radiology department of HEGP (only unblinded center) will have the knowledge of the trial arm.
  Patient will be blinded from randomization arm using headphones and/or virtual headset.
  The research personnel will be trained accordingly and will keep a separate file with patient's images to ensure that they are not transferred on the Pacs system (Carestream).
  The research assistant will discard the products after completion of the procedure in specific containers, that will not be accessible to the patient or to nurses and technicians directly involved in the current patient's care.
  Patient's blindness will be assessed using a blinding index after GAE and at the 3-month follow-up visit. The proposed blinding index is scaled to an interval of -1 to 1, 1 being complete lack of blinding, 0 being consistent with perfect blinding and -1 indicating opposite guessing which may be related to unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization group (Experimental): Genicular arteries embolization of the target knee will be performed using an ethiodized oil-based emulsion (3:1 mix of ethiodized oil and contrast agent ioversol 300 mgI/ml); 86 patients will be allocated to embolization group (2:1 randomization).
  Interventions: Drug: Ethiodized Oil-based emulsion
- Sham group (Sham Comparator): All the gestures will be mimed using the same equipment as in GAE group. Superficial femoral artery catheterization, selective catheterization of target arteries and emulsion injection will be mimicked by the interventional radiologist (table movements, syringes manipulation) to keep the patient blind from the actual treatment.
  44 patients will be allocated to sham group (2:1 randomization).
  Interventions: Procedure: Sham-operation

INTERVENTIONS:
Drug: Ethiodized Oil-based emulsion — Embolization of genicular arteries
  Arms: Embolization group
Procedure: Sham-operation — Mimicked catheterization and embolization of genicular arteries
  Arms: Sham group

SUMMARY:
Knee OsteoArthritis (KOA) is a common disease associated with pain and impaired function. Many patients are not relieved of their symptoms with enough efficacy by conservative treatments. Genicular Arteries Embolization (GAE) is a new minimally invasive endovascular treatment allowing symptoms relief. The investigator previously demonstrated the safety of GAE using an ethiodized oil-based emulsion for the treatment of painful knee osteoarthritis in a first-in-man single-arm clinical trial called LipioJoint-1 (clinicaltrials.gov: NCT04733092; EUDRACT: 2020-002206-10). This phase 1 study also provided encouraging evidence of GAE efficacy on knee pain and function.

The purpose of LipioJoint-2 study is to assess GAE efficacy using an ethiodized oil-based emulsion for the treatment of painful knee osteoarthritis in a multicenter, prospective, randomized sham-controlled clinical trial.

DETAILED DESCRIPTION:
Patients will be screened during current practice consultation in each recruiting center (Screening Visit). When a patient will meet the eligibility criteria, he will be informed about the protocol.

The Interventional Radiologist will further explain the protocol to the patient and check inclusion/non-inclusion criteria during baseline visit. The date of signature of the informed consent by the patient will be considered as the date of inclusion. GAE (embolization) will be scheduled within the next few days.

Randomization will occur during the embolization visit, before patient is taken to the operating room. Randomization in a 2:1 ratio of GAE using emulsion to the sham procedure will be performed with stratification on Kellgren and Lawrence score (2-3 versus 4). All target arteries will be injected with an ethiodized oil-based emulsion (GAE group). Patient will be kept blind to the actual treatment using headphones or virtual headset.

Follow-up visits will be scheduled 1, 3, 6 and 12 months after randomization. Patient will be informed about his randomisation group (GAE or sham) after the completion of questionnaires (VAS pain, WOMAC, EQ-5D, HAD) at the 3-month visit and will be allowed to choose further medical & clinical management of his target KOA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary KOA according to the classification of the American College of Rheumatology (ACR) (5)
* Radiographic Kellgren and Lawrence score ≥ 2 (6)
* VAS pain score ≥ 40 mm (scale 0-100 mm)
* Previous intra-articular injection in the target knee
* Patient not eligible to knee surgery
* For woman of childbearing potential: negative bêta-HCG before randomization
* Social security affiliation
* Signed informed consent
* Good understanding of the French language

Exclusion Criteria:

* Intra-articular injection of any product in the target joint within 3 months before embolization
* Prior knee surgery other than ligament repair
* Any inflammatory joint disease other than osteoarthritis
* Any contra-indication to puncture of the ipsilateral femoral artery
* Current treatment with cyclosporine, tacrolimus, cisplatine, vancomycine, amphotericine B or any aminoside
* Ipsilateral symptomatic hip OA
* Treated hyperthyroidism
* Known severe allergy to Lipiodol® and/or iodine contrast medium
* Known moderate to severe kidney failure (creatinine clearance < 30 45 ml/min)
* Known right-to-left cardiac shunt or intra-tumoral vascular shunt
* Asthma attack in the 8 days before randomization
* Exploration or treatment with radioactive iodine scheduled within 1 month after randomization
* Symptomatic atheromatous lesion in the ipsilateral limb
* Patient unable or unwilling to comply with the follow-up schedule (at the investigator's discretion)
* Vulnerable populations (such as pregnant or breastfeeding women, patient under guardianship curatorship, deprived of liberty)
* Patient under exclusion period in another trial
* Patient on AME (state medical aid)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of pain assessed by a Visual Analogue Scale (VAS) at 3 months compared to randomization. | 3 months
  VAS pain is a validated, self-reported instrument assessing average pain over the past 48 hour period. Score ranges from 0 (no pain) to 100 (worst possible pain).

SECONDARY OUTCOMES:
Change of pain assessed by a Visual Analogue Scale (VAS) at 1 month compared to randomization. | 1 month
  VAS pain is a validated, self-reported instrument assessing average pain over the past 48 hour period. Score ranges from 0 (no pain) to 100 (worst possible pain).
Change of pain assessed by a Visual Analogue Scale (VAS) at 6 months compared to randomization. | 6 months
  VAS pain is a validated, self-reported instrument assessing average pain over the past 48 hour period. Score ranges from 0 (no pain) to 100 (worst possible pain).
Change of pain assessed by a Visual Analogue Scale (VAS) at 12 months compared to randomization. | 12 months
  VAS pain is a validated, self-reported instrument assessing average pain over the past 48 hour period. Score ranges from 0 (no pain) to 100 (worst possible pain).
Change of the patient's global assessment of her/his health measured by the Visual Analogue Scale of EQ-5D questionnaire (EQ VAS) at 1, 3, 6, 12 months compared to randomization. | Up to 12 months
  EQ-5D questionnaire is a validated, self-reported instrument assessing "today" health-related quality of life. EQ VAS is the second part of EQ-5D, consisting in a Visual Analogue Scale of health. Score ranges from 0 (worst health) to 100 (best health).
Change of the Western Ontario and McMaster Universities Arthritis (WOMAC) total and sub-scores (pain, function,stiffness) at 1, 3, 6, 12 months compared to randomization. | Up to 12 months
  WOMAC questionnaire is a validated, self-reported instrument assessing the daily condition of patients with osteoarthritis of the lower limb. It has a multidimensional scale comprising 24 items grouped into three dimensions: pain (5 items), stiffness (2 items), and physical functioning (17 items).
  Likert scale will be normalized to 100. Scores ranges from 0 (no impairment) to 100 (severe impairment).
Change of the Knee injury and Osteoarthritis Outcome Score (KOOS) total and sub-scores at 3 months compared to randomization. | 3 months
  KOOS questionnaire is a validated, self-reported instrument assessing the daily condition of patients with osteoarthritis of the lower limb. It has a multidimensional scale comprising 42 items grouped into five dimensions: pain (9 items), symptoms (7 items), activities of daily living function (17 items), sport and recreation function (5 items), quality of life (4 items).
  A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included.
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic assessment scales and generic measures.
Change of the Hospital Anxiety and Depression (HAD) score and sub-scores at 3 months compared to randomization. | 3 months
  HAD questionnaire is a validated, self-reported instrument assessing the levels of anxiety and depression. It has a multidimensional scale comprising 14 items grouped into two dimensions: anxiety (7 items), and depression (7 items). Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. Total score ranges from 0 (no impairment) to 42 (severe impairement). A total sub-scale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Change of semi-quantitative MRI scoring at 6 months compared to randomization. | 6 months
  Semi-quantitative MRI scoring may include Whole-Organ Magnetic Resonance Imaging Score (WORMS), Knee Osteoarthritis Scoring System (KOSS), Boston-Leeds Osteoarthritis Knee Scoring (BLOKS), MRI Osteoarthritis Knee Score (MOAKS).
Description of pain medication at Month 1, 3, 6, 12. | Up to 12 months
  Pain medication will be described using analgesic level.
Description of non-pharmacological treatments for target knee in both groups at 1, 3, 6, and 12 months. | Up to 12 months
  Non-pharmacological interventions may include, but are not limited to, physiotherapy, osteopathy, acupuncture, massage, electroanalgesia, laser therapy, low-level light therapy, meditation.
Number of responder patients under OMERACT-OARSI definition in both groups at 3, 6 and 12 months. | Up to 12 months
  A patient is defined as responder under OMERACT-OARSI criteria if one of the following conditions is satisfied:
  * Improvement in pain (0-100 mm VAS) or in WOMAC function score ≥50% and absolute change ≥20 is observed or
  * Improvement in at least 2 of the 3 following conditions:
    * Pain (0-100 mm VAS) ≥20% and absolute change ≥10
    * WOMAC function score ≥20% and absolute change ≥10
    * Patient's global assessment of her/his health (0-100 mm EQ-5D VAS) ≥20% and absolute change ≥10
Number of patients reaching an acceptable symptom state (PASS) in both groups at 3, 6, and 12 months. | Up to 12 months
  PASS is defined for each patient reported outcome as:
  * Pain (0-100 mm VAS) ≤32.3,
  * Patients global assessment of her/his health (0-100 mm EQ-5D VAS) ≤32,
  * WOMAC function score (0-100) ≤31.
Number and description of adverse events and serious adverse events at 1, 3, 6 and 12 months. | Up to 12 months
  Adverse events are defined according to Article 2 of the Regulation (EU) No 536/2014. Intensity of adverse events will be graded using Clavien-Dindo classification and CTCAE v 5.0.
Description of target knee events in both groups at 6 and 12 months. | Up to 12 months
  Events of interest includes intra-articular injections, embolization, surgery.
Incremental efficiency of genicular arteries embolization compared to sham treatment (medico-economic analysis). | 6 months
  Medico-economic study: incremental cost utility ratio

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAPOVAL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Saint Antoine - APHP, Paris
  - Hôpital Cochin - APHP, Paris
  - Hôpital européen Georges Pomidou - APHP, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).